CLINICAL TRIAL: NCT02893436
Title: Time Prediction for Complete Recovery From Neuromuscular Blockade After Visual Recovery With Double Burst Stimulation
Acronym: DBS PREDICTION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2014/DBSPREDICTION-SCHMARTZ
Record Dates: First submitted 2016-08-31; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-08

CONDITIONS: Anesthesia; Surgery
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Curarized patients
  Interventions: Procedure: Surgery with tracheal intubation curarisation

INTERVENTIONS:
Procedure: Surgery with tracheal intubation curarisation

SUMMARY:
The purpose is to calculate the time for an optimal recovery (T4/T1 > 0.9) from the moment when 2 responses to double burst stimulation are visually identical and this for 95% of patients.

DETAILED DESCRIPTION:
Neuromuscular monitoring is a basic monitoring for all curarised patients. Acceleromiography is used to supervise neuromuscular blockade and allow measuring in an objective and quantitative manner the curarisation level during surgery and phase of recovery from neuromuscular blockade. Various parameters are usually measured during surgery:

* T4/T1 ratio: ratio between the 4th and 1st response to "train of four" stimulation (TOF, 4 stimulations of 0.2 ms in 2 s). Neuromuscular recovery is considered appropriate if T4/T1 ratio is > 0.9
* Double burst stimulation (DBS): 2 short tetanic stimulations separated by an interval of 750 ms.

It is known that when DBSs induce the same visual and/or tactile response, T4/T1 recovery time is > 0.6. However, for an optimal recovery, T4/T1 ratio must be > 0.9.

This study will analyze the interval between the moment when DBSs are visually identical and the T4/T1 ratio is > 0.9, from anesthesia sheet of patients undergone surgery with tracheal intubation curarisation.

Results will define a minimum time to have an optimal recovery after having visually identical DBS responses.

ELIGIBILITY:
Inclusion Criteria:

* ASA score 1-3
* Needing a surgery with tracheal intubation curarisation

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient curarised at Nancy Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Time interval between the moment when DBSs are visually identical and the T4/T1 ratio is > 0.9 | day 0
  measured with TOF-Watch Sx

CONTACTS AND LOCATIONS:
Overall Officials: Denis Schmartz, Principal Investigator — CHRU Nancy, France
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided